CLINICAL TRIAL: NCT06061120
Title: Non-invasive Differentiation of Supraventricular Tachyarrhythmias by Questionnaire and High-resolution ECG in the Context of Ablation Treatment
Brief Title: Non-invasive Differentiation of Supraventricular Tachyarrhythmia
Acronym: NIDSA
Status: Recruiting | Type: Observational
Sponsor: RWTH Aachen University (Other)
Collaborators: Department of Internal Medicine I - Cardiology (Unknown); KKS -Kardiologisches Klinisches Studienzentrum (Unknown); Chair of Medical Information Technology Helmholtz Institute, RWTH Aachen University (Unknown)
Responsible Party: Principal Investigator, Matthias Zink, Dr. med., RWTH Aachen University
Other Study IDs: CTCA 21-083
Record Dates: First submitted 2022-10-25; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Supraventricular Arrhythmia; Atrial Fibrillation
Keywords: Electrocardiogram; Signal-averaged P-Wave; Questionnaire; Supraventricular Arrhythmia; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Questionnaire - Supraventricular arrhythmia: Questionnaire about triggers and stops of supra ventricular arrhythmia
- Extended ECG - Effect of electrophysiological ablation: Extended signal-averaged ECGs in patients with ablation of supra ventricular ablation
  Interventions: Device: Recording of an extended high-resolution ECG
- Extended ECG - Virtual atrial Electrocardiogram: Improve visualisation of atrial arrhythmia by means of extended signal-averaged ECGs
  Interventions: Device: Recording of an extended high-resolution ECG

INTERVENTIONS:
Device: Recording of an extended high-resolution ECG — Recording of an extended high-resolution ECG
  Groups: Extended ECG - Effect of electrophysiological ablation; Extended ECG - Virtual atrial Electrocardiogram

SUMMARY:
1. Questionnaire for supraventricular tachycardia: About history and targeted diagnosis of supraventricular tachycardia
2. Extended Signal-averaged ECG for detailed P-Wave analysis and to calculate a virtual atrial electrocardiogram (ECG)

DETAILED DESCRIPTION:
1. Questionnaire Patient questionnaires on supraventricular tachycardia including atrial fibrillation often refer to the symptoms of the cardiac arrhythmia and the resulting limitations in everyday life. The evaluation of these questionnaires only allows a rough differentiation between the various cardiac arrhythmias. Nevertheless, it is known that supraventricular tachycardias are influenced by the sympathetic and parasympathetic nervous system. For example, tachyarrhythmias can begin or be terminated with a reentry circuit through the atrioventricular (AV) node by Valsalva manoeuvres or some other change in tone of the nervus vagus. For atrioventricular reentrytachycardia (AVNRT) in particular, an increased probability of occurrence in poststress phases has been described, as well as an association with certain behaviours such as positional changes, but also alcohol and drug consumption. To date, there is no systematic questionnaire on the specific triggering and terminating components. All patients referred for ablation of a supraventricular arrhythmia and potentially included in this project will receive a detailed history of the triggering and terminating factors using a structured questionnaire, as well as two validated supraventricular tachycardia questionnaires (5Q-3L and ASTA) to classify the results of our questionnaire.
2. Extended ECG A high-resolution and signal-averaged ECG is recorded with a significantly higher resolution than a 12-lead ECG over a period of several minutes. Additional electrode positions are also used in the vicinity of the examined structure, e.g. the left atrium. The signal from several recorded heartbeats is then averaged. This preserves repetitive smallest atrial excitation patterns and changes. In this way, it is possible to find indications of cardiac arrhythmias like atrial fibrillation in the signal-averaged ECG, which were not detectable in a 12-lead ECG.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for ablation of a supraventricular tachycardia (atrial fibrillation, typical atrial flutter, AV nodal reentry tachycardia, accessory pathway)
* majority

Exclusion Criteria:

* Unstable patient with need for intensive medical care
* Lack of language skills or limited cognitive abilities that prevent a differentiated anamnesis and information.

Exclusion criteria for study section Questionnaire:

- Competing clinically present arrhythmias, including relevant supra- and ventricular extrasystole (>5%/die).

Exclusion criteria for study section Extended high-resolution ECG:

* Previous electrophysiological ablation at the same site for atrial fibrillation.
* Relevant supra- and ventricular extrasystole (>5%/die).
* Other clinically present arrhythmias are not excluded if they can be sequentially triggered and ablated (e.g. atrial fibrillation and atrial flutter). Since separate detection is possible with the high-resolution ECG.
* Implanted active electrical device (e.g. pacemaker, defibrillator, deep brain pacemaker)
* Allergy to measuring electrodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort for study section Questionnaire: 1000 evaluable questionnaires are targeted. Every suitable potential respondent will be invited and interviewed during the data collection period. After 400 subjects in the questionnaire section, an interim evaluation will be carried out.
  Cohort for study section extended high-resolution ECG: In a feasibility study, signal-enhanced ECGs will be recorded in a subgroup of cohort before, during and after ablation with the aim of non-invasive ECG diagnostics. There are no published empirical values for this and 250 subjects will be notified. After 100 subjects in the high-resolution ECG section, an interim evaluation will be carried out.
Sampling Method: Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Triggers of supraventricular arrhythmia | 2 years
  Anamnestic and ECG measured triggers of supra ventricular arrhythmia

SECONDARY OUTCOMES:
P-Wave duration | 2 years
  Characteristics and changes by ablation of atrial electrical activation will be analyzed by means of signal-averaged P-Wave parameters
P-Wave amplitude | 2 years
  Characteristics and changes by ablation of atrial electrical activation will be analyzed by means of signal-averaged P-Wave parameters
P-Wave PQ time (time mesaured from begin of P-wave to begin of Q-Peak) | 2 years
  Characteristics and changes by ablation of atrial electrical activation will be analyzed by means of signal-averaged P-Wave parameters
Signal-averaged P-Wave sample entropy | 2 years
  Characteristics and changes by ablation of atrial electrical activation will be analyzed by means of signal-averaged P-Wave parameters
Signal-averaged P-Wave shannon entropy | 2 years
  Characteristics and changes by ablation of atrial electrical activation will be analyzed by means of signal-averaged P-Wave parameters
Signal-averaged P-Wave complexity | 2 years
  Characteristics and changes by ablation of atrial electrical activation will be analyzed by means of signal-averaged P-Wave parameters
Visualisation of a signal-averaged P-Wave before and after catheter ablation with qualitative review of morphology | 2 years
  By recording of unfiltered high-resolution ECG and calculation of a signal-averaged P-Wave and other post-processing techniques a better visualization of ongoing arrhythmia shall be achieved

CONTACTS AND LOCATIONS:
Overall Officials: Matthias D Zink, MD, Principal Investigator — RWTH Aachen University
Locations (1):
- RWTH Aachen University, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared on reasonable request after data is already published
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Derived] Fantazi N, Hermans BJM, Zeemering S, Berbers J, Emrani M, Napp A, Marx N, Gramlich M, Schotten U, Zink MD. Acute effect of cryoballoon pulmonary vein isolation on the signal-averaged P-wave. Front Cardiovasc Med. 2026 Jan 20;12:1728939. doi: 10.3389/fcvm.2025.1728939. eCollection 2025. PMID 41640583